CLINICAL TRIAL: NCT01034124
Title: Mechanisms Underlying Drug-Diet Interactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Mary F. Paine, The University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UNC-CH 05-2951
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Pharmacokinetics
Keywords: warfarin; midazolam; cranberry juice; pharmacokinetics
MeSH Terms: interventions — Warfarin; Vitamin K; Midazolam; Vitamin K 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water (Placebo Comparator)
  Interventions: Drug: warfarin, vitamin K, midazolam
- Cranberry juice (Active Comparator)
  Interventions: Drug: warfarin, vitamin K, midazolam

INTERVENTIONS:
Drug: warfarin, vitamin K, midazolam — warfarin tablet single dose (10 mg) vitamin K tablet single dose (10 mg) midazolam syrup single dose (5 mg)
  Other Names: Coumadin; Mephyton; Versed

SUMMARY:
Similar to the well publicized "grapefruit juice effect", ongoing studies are evaluating the interaction potential of other dietary substances on drug disposition. This study is designed to determine whether the mechanism underlying the enhancement of the anticoagulative effect of warfarin by cranberry juice is due to inhibition of warfarin metabolism by the juice. A secondary objective is to determine whether cranberry juice elicits a grapefruit juice-type interaction with midazolam.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Healthy
* Not taking medications known to modulate CYP2C9 and CYP3A activity
* Able to understand the consent process

Exclusion Criteria:

* Allergy to cranberry products, warfarin, vitamin K, or midazolam
* Pregnant or breast-feeding women
* Baseline INR >1.2
* History of significant medical conditions that could increase risk
* Concomitant medications known to modulate CYP2C9 and CYP3A activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
AUC | 0-96 hr

SECONDARY OUTCOMES:
Cmax | varies

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Paine, Ph.D., Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC-Chapel Hill General Clinical Research Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Ngo N, Yan Z, Graf TN, Carrizosa DR, Kashuba AD, Dees EC, Oberlies NH, Paine MF. Identification of a cranberry juice product that inhibits enteric CYP3A-mediated first-pass metabolism in humans. Drug Metab Dispos. 2009 Mar;37(3):514-22. doi: 10.1124/dmd.108.024968. Epub 2008 Dec 29. PMID 19114462